CLINICAL TRIAL: NCT03238534
Title: Relief of Heartburn and Epigastric Pain Comparing Neobianacid® With Omeprazole: a Randomized, Double Blind, Double Dummy, Reference Product Controlled, Parallel Group, Non-inferiority Clinical Study
Brief Title: Efficacy and Safety Evaluation of Neobianacid® in GERD and EPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Doppel Farmaceutici (Unknown); University of Roma La Sapienza (Other); BMR Genomics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABO-NB-15
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2021-12

CONDITIONS: GERD; EPS
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind (patient+investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole 20mg (Active Comparator): Patients will be provided with enough amount of 20 mg omeprazole [30' before meal] and Neobianacid® placebo [30' after meal] (both per os) to complete the first phase of the treatment (day 1-27). Then, at day 28, the patients will be provided with Neobianacid® that can be administered on demand until the study end (day 56). Malgradate will be also provided as rescue medication.
  Treatment regimen:
  Day 0-13 Breakfast: Omeprazole + Neobianacid® placebo; Lunch: Neobianacid® placebo; Midafternoon: Neobianacid® placebo; Dinner: Neobianacid® placebo; Before going to bed: Neobianacid® placebo.
  Day14-27 Breakfast: Omeprazole+ Neobianacid® placebo on demand Lunch: Neobianacid® placebo on demand Dinner: Neobianacid® placebo on demand Any other time: Neobianacid® placebo on demand, if needed
  Day28-55 Breakfast: Neobianacid® on demand Lunch: Neobianacid® on demand Dinner: Neobianacid® on demand Any other time: Neobianacid® on demand, if needed
  Interventions: Drug: Omeprazole 20mg; Other: Neobianacid® placebo
- Neobianacid® (Experimental): Patients will be provided with enough amount of Omeprazole placebo [30' before meal] and Neobianacid® [30' after meal] (both per os) to complete the first phase of the treatment (day 1-27). Then, at day 28, the patients will be provided with Neobianacid® that can be administered on demand until the study end (day 56). Malgradate will be also provided as rescue medication.
  Treatment regimen:
  Day 0-13 Breakfast: Omeprazole placebo + Neobianacid® Lunch: Neobianacid® Midafternoon: Neobianacid® Dinner: Neobianacid® Before going to bed: Neobianacid®
  Day14-27 Breakfast: Omeprazole placebo + Neobianacid® on demand Lunch: Neobianacid® on demand Dinner: Neobianacid® on demand Any other time: Neobianacid® on demand, if needed
  Day28-55 Breakfast: Neobianacid® on demand Lunch: Neobianacid® on demand Dinner: Neobianacid® on demand Any other time: Neobianacid® on demand, if needed
  Interventions: Device: Neobianacid®; Other: Omeprazole placebo

INTERVENTIONS:
Device: Neobianacid® — Oral administrations of Neobianacid® (30' after meals and on demand)
  Arms: Neobianacid®
Drug: Omeprazole 20mg — Daily administration Omeprazole 20mg (per os, 30' before breakfast).
  Arms: Omeprazole 20mg
Other: Neobianacid® placebo — Oral administrations of Neobianacid® placebo (30' after meals and on demand)
  Arms: Omeprazole 20mg
Other: Omeprazole placebo — Daily administration Omeprazole placebo (per os, 30' before breakfast).
  Arms: Neobianacid®

SUMMARY:
Comparison of Neobianacid® clinical efficacy to omeprazole in relief of heartburn or epigastric pain

DETAILED DESCRIPTION:
Comparison of heartburn or epigastric pain severity following administration of Neobianacid® (Group B) or omeprazole (Group A) from day 0 to day 27. An ad-hoc placebo will be also administered in both treatment arms. Then, a following phase (day 28-55) will follows in which Neobianacid® will be administered (on demand) to both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 - 70 years old (inclusive).
2. Patients presenting one or both the 2 following conditions:

   * Patients presenting heartburn who have been already diagnosed with uncomplicated gastroesophageal reflux disease (GERD) or whose symptoms are consistent with a clinical diagnosis of uncomplicated GERD.
   * Patients who have been already diagnosed with uncomplicated Epigastric Pain Syndrome (EPS) or whose symptoms are consistent with a clinical diagnosis of uncomplicated EPS according to Rome III criteria.
3. A gastroscopy is to be performed if not already performed during the previous 3 years and the symptomatology is unchanged.
4. Patients having a VAS score ≥ 30mm and ≤ 70mm (VAS related to heartburn/ epigastric pain) for at least 6 out of 14 days preceding the screening visit.
5. Postmenopausal women i.e. women who have not experienced a menstrual bleed for a minimum of 12 months or women who have undergone surgical sterilization (tubal closure or ovaries removal). Otherwise, necessity for women of childbearing potential to follow a reliable contraceptive treatment.
6. Ability of the patients (in the Investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects.
7. Patients who agree not to alter their diet in any way for the duration of the trial and to maintain it at steady state.
8. Patients who agree not to make any major lifestyle changes during the trial.
9. Consent to the study and willing to comply with all its procedures.
10. Chronic therapies (if not related to the gastroenterological pathologies object of the study, according to the opinion of Investigator) are allowed, if the regimen is maintained stable during the whole study.

Exclusion Criteria:

1. Patients with heartburn/epigastric pain who have not previously responded to antacid or PPI.
2. Patients having a VAS score > 70mm (VAS related to heartburn/ epigastric pain) for at least 6 out of 14 days preceding the screening visit.
3. Patient presenting one of the following condition:

   1. anemia;
   2. chronic gastrointestinal bleeding;
   3. antibiotic use, including antifungal and antimalarial medication within 2 months preceding the start of the study;
   4. progressive unintentional weight loss;
   5. persistent or recurrent vomiting;
   6. epigastric mass;
   7. acute episode with dyspnea, diaphoresis, or tachycardia;
   8. anorexia;
   9. nausea or vomiting;
   10. dysphagia or odynophagia.
4. Patients under triple therapy or eradication therapy against Helicobacter pylori.
5. Patients using any drugs that could affect symptoms, such as NSAIDS, antacids, anti- secretory agents including proton pump inhibitors (other than the study products) and histamine H2-receptor antagonists or prokinetic or antiulcer agents, gastric mucosal protectants, anticholinergics and/or cholinergic agents. Moreover, the patients will be asked to avoid any drugs of the above mentioned since the beginning of the study (since pre-screening visit) until the end of the study.
6. Patients with the presence of the following conditions: erosive GERD, Barrett's oesophagus or oesophageal stricture, active or healing gastroduodenal ulcer (except scars) or any other GI disease, which is not mentioned in the inclusion criteria; history of gastric, duodenal or esophageal surgery; malignant disease of any kind; gallstone. Any chronic disease that may affect the gastrointestinal upper tract.
7. Patients with clinically significant liver disease (AST/SGOT, ALT/SGPT >2 upper limits of normal).
8. Patients with clinically significant renal disease (serum creatinine >1.5 mg/dl).
9. Patient having any other conditions or disease that the Investigator will consider non-appropriate to the study (any severe disease of another major body system other than GI tract).
10. Patients with porphyria, hypophosphatemia, cachexia.
11. Pregnant or nursing women or women planning to become pregnant during the study.
12. Patients with a history of alcohol or drug abuse.
13. Known hypersensitivity or intolerance to any components of the study products or rescue medication.
14. Subjects presenting contraindications to the study products or rescue medication, according to concerning Summaries of Product Characteristics (SPC), e.g. for omeprazole, patients suffering from rare hereditary problems of fructose intolerance, Glucose Galactose Malabsorption (GGM) or sucrase-isomaltase deficiency.
15. Patients being treated with any drug whose pharmacokinetics can interfere with the intake of omeprazole or magaldrate (e.g., for omeprazole, the active substances known as CYP2C19 or CYP3A4 inhibitors, as clarithromycin and voriconazole, or inductors, as rifampicin and St. John's wort, Hypericum, or both) or with any drug with which omeprazole, neobianacid or magaldrate are able to interact.
16. Patient participating to any investigational drug trial within 4 weeks before screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Heartburn or epigastric pain severity through treatment (Day-1 to Day13) | Day-1 to Day13
  Comparison of heartburn or epigastric pain severity by means of a 100mm VAS scale (from "no symptoms" to "overwhelming symptoms"); from Baseline to Day 13, between groups. Baseline is defined as Day -1

SECONDARY OUTCOMES:
Heartburn or epigastric pain severity through treatment (Day-1 to Day7) | Day-1 to Day7
  Comparison of heartburn or epigastric pain severity by means of a 100mm VAS scale (from "no symptoms" to "overwhelming symptoms") from Baseline to Day 1, Day 3 and Day 7, between groups
Heartburn or epigastric pain severity through treatment (Day14 to Day27) | Day14 to Day27
  Assessment of heartburn or epigastric pain severity by means of a 100mm VAS scale (from "no symptoms" to "overwhelming symptoms"); from Day 14 to Day 27 between groups.
Assessment of of rescue medication use | Day-1 to Day55
  Assessment of use (starting date and quantity) of rescue medication (antacid); from Baseline to Day 13, from Day 14 to Day 27 and from Day 28 to Day 55, between groups.
Tablets of Neobianacid® Vs. Neobianacid® placebo Day14 to Day27 | Day14 to Day27
  Assessment of number of tablets of Neobianacid® on demand in comparison to Neobianacid® placebo on demand; from Day 14 to Day 27, between groups.
Tablets of Neobianacid® Vs. Neobianacid® placebo Day28 to Day55 | Day28 to Day55
  Assessment of number of tablets of Neobianacid® on demand; from Day 28 to Day 55, between groups.
Improvement in symptomatology | Day-1 to Day56
  Improvement in symptomatology, by means of Gastrointestinal Symptom Rating Scale Questionnaire - GSRS; Day 14, Day 28 and Day 56 versus Baseline, between groups.
Improvement in quality of life | Day-1 to Day56
  Improvement in quality of life, by means of Gastrointestinal Quality of Life Index - GIQLI questionnaire; Day 14, Day 28 and Day 56 versus Baseline, between groups.
Evaluation of treatment | Day-1 to Day56
  Evaluation of treatment by means of Overall Treatment Evaluation - OTE; Day 14, 28 and 56, between groups.

OTHER OUTCOMES:
intestinal microbiota characterization | Day-1 and Day28
  Characterization of the whole intestinal microbiota carried out by means of the analysis of faecal samples; Baseline and Day 28.

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Azienda Ospedaliera Santa Maria Goretti, Latina, Rome
  - Ospedale Civile San Salvatore, L’Aquila
  - Policlinico San Matteo Pavia Fondazione IRCCS, Pavia
  - Azienda Ospedaliera Perugia, Perugia
  - Azienda Ospedaliera Sant'Andrea, Rome
  - Ospedale San Giovanni Addolorata, Rome
  - Ospedale Sandro Pertini, Rome
  - Ospedale Sant'Eugenio, Rome
  - Policlinico Umberto I, Rome
  - Policlinico Universitario A. Gemelli, Rome
  - Policlinico Universitario Campus Biomedico di Roma, Rome
  - Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi d'Aragona, Salerno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corazziari ES, Gasbarrini A, D'Alba L, D'Ovidio V, Riggio O, Passaretti S, Annibale B, Cicala M, Repici A, Bassotti G, Ciacci C, Di Sabatino A, Neri M, Bragazzi MC, Ribichini E, Radocchia G, Iovino P, Marazzato M, Schippa S, Badiali D. Poliprotect vs Omeprazole in the Relief of Heartburn, Epigastric Pain, and Burning in Patients Without Erosive Esophagitis and Gastroduodenal Lesions: A Randomized, Controlled Trial. Am J Gastroenterol. 2023 Nov 1;118(11):2014-2024. doi: 10.14309/ajg.0000000000002360. Epub 2023 Jun 13. PMID 37307528